CLINICAL TRIAL: NCT06992908
Title: Reliability of Artificial Intelligence for Treatment Decision Recommendation for Adult Skeletal Open Bite Patients: A Diagnostic Accuracy Pilot Study
Brief Title: Reliability of Artificial Intelligence for Treatment Decision for Adult Skeletal Open Bite Patients
Acronym: AIASOBP
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Saeed Abdullah Saeed Badyah, Master's student., Cairo University
Other Study IDs: Adult skeletal open bite cases; Self-funded by me. (Other: Self-funded by me.)
Record Dates: First submitted 2025-04-24; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Openbite; Artifical Intelligence
MeSH Terms: conditions — Open Bite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: MLG acts as learning group.: Cephalometric readings parameters of cases with their decisions will be used in this group for training the machine to be able to make a decision.
- Group 2: TG acts as a test group: The programmer will put parameters as input and then ask the AI model to decide on an output of the model, either camouflage or surgery.

SUMMARY:
This study evaluated a specially designed AI model developed by a programmer using x-ray readings and corresponding treatment decisions from 70% of the cases (either orthodontic treatment only or orthodontic treatment with surgery).

For the evaluation, we will use the remaining 30% of cases. "Subsequently, to assess its performance, the model was tested on the remaining 30% of cases. The programmer provided only the X-ray readings as input. The AI model was then tasked with classifying.

DETAILED DESCRIPTION:
In this study, all patients were treated completely with a well-finished result by expert orthodontists. This study evaluates whether an artificial intelligence (AI) model can enhance treatment decisions for adult skeletal open bite cases by predicting the optimal intervention, either orthognathic surgery or camouflage, using cephalometric readings as input data.

First, a total of 53 cases were analyzed, which were divided into two groups:

70% were allocated to the machine learning group (MLG), while the remaining 30% constituted the test group (TG). Cephalometric analysis for all patients was performed using Dolphin Imaging 11.5 Premium software, along with determining the appropriate treatment decision, either camouflage or orthognathic surgery.

The data obtained from MLG serves as training data for the AI model to classify cases based on their cephalometric data, whether for camouflage or orthognathic surgery. The input data consisted of cephalometric readings along with a decision.

Second, after machine learning, validation takes place to examine the ability of the machine to make decisions through some cases from MLG.

The third step will evaluate the machine's ability to accurately determine case decisions based on cephalometric readings. The results produced by the machine will be compared to the actual decisions made, as all these cases were treated under the supervision of orthodontic professors.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Adult patients with anterior skeletal open bite (at least 3mm opening)
* Completed their treatment successfully.
* Well-documented cases with comprehensive preoperative and postoperative lateral cephalometric x-rays were considered.

Exclusion Criteria:

* Patient below 18 years.
* Improperly finished orthodontic treatment.
* Incomplete documentation.
* cleft lip and palate patient, patient with syndromes.
* Dental open bite.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult anterior skeletal open bite patients with at least 3mm opening.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2024-05-12 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
accuracy of diagnostic test | through study completion, an average of 1 year".
  In this study, the investigators have only one outcome, which is the accuracy of a diagnostic test.
  This test is based on the comparison of the results of machine learning decisions with a conventional method, which is an expert orthodontist's decision.
  Accuracy = (true positives + true negatives) / (total) A true positive will be the correct prediction of camouflage. A true negative will be the correct prediction of orthognathic surgery. Total means the total test set cases. All cases are randomly distributed. The investigators use the skeletal and dental cephalometrical parameters , some of which are angles measured by degrees, and others are linear measurements measured by millimeters.
  SNA SNB ANB SN/PP SN/MP Maxillary-mandibular plane angle Anterior facial height Posterior facial height Jarabak ratio Gonial angle Lower anterior facial height Open bite Maxillary anterior teeth inclination Mandibular anterior teeth inclination

CONTACTS AND LOCATIONS:
Overall Officials: Dina Osman, Associate Professor, Study Director — supervisor; Mostafa El-Dawlatly, Associate Professor, Study Director — supervisor
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No